CLINICAL TRIAL: NCT06297291
Title: The Global Paradise® System US Post Approval Study (US GPS)
Brief Title: Global Paradise System US Post Approval Study
Acronym: US GPS
Status: Recruiting | Type: Observational
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN 0984
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
Keywords: Blood Pressure; Uncontrolled Hypertension; Essential Hypertension; Resistant Hypertension; Renal Denervation; Ultrasound Renal Denervation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Prospective Ultrasound Renal Denervation Treatment: Hypertension patients that meet the eligibility criteria for treatment with Recor Medical Paradise Ultrasound Renal Denervation System will be enrolled and followed post-procedure for 5 years.
  Interventions: Device: Paradise Ultrasound Renal Denervation Treatment
- RADIANCE CAP Transfer: Subjects enrolled in the RADIANCE Continued Access Protocol (CAP) study that are still active and have already completed their post-procedure 12-month follow-up visit are invited to participate in US GPS for long-term annual follow-up visits. These subjects will have already received the ultrasound Renal Denervation treatment under the RADIANCE CAP protocol and will not receive the procedure under the US GPS protocol.

INTERVENTIONS:
Device: Paradise Ultrasound Renal Denervation Treatment — The Paradise Ultrasound Renal Denervation System (Paradise Ultrasound RDN) is an FDA-approved catheter-based system to treat hypertension by ablating the nerves around the renal arteries, disrupting the overactive sympathetic nerves that can cause high blood pressure. The Paradise procedure uses ultrasound energy to calm the nerves near the kidneys to help lower blood pressure.
  Treatment is usually done in an outpatient setting and typically takes about an hour to perform. As a part of the treatment, a small flexible tube (catheter) is guided into the blood vessels near the kidneys and 7 seconds of ultrasound energy is applied 2-3 times. Both sides are treated and then the catheter is removed, leaving nothing behind. After the procedure, some people go home the same day or some stay overnight.
  Other Names: Paradise Ultrasound RDN
  Groups: Prospective Ultrasound Renal Denervation Treatment

SUMMARY:
The objective of the Global Paradise® System US Post Approval Study (US GPS) is to evaluate the real-world use of the Paradise Ultrasound Renal Denervation System indicated for patients who are unable to lower their blood pressure with lifestyle changes and medication. This system is comprised of a catheter, cable, balloon, and generator and has received FDA approval in the United States. Information collected in this study will be analyzed to better understand the long-term safety and effectiveness of treatment with the Paradise System for patients with high blood pressure.

DETAILED DESCRIPTION:
In some patients with high blood pressure, the nerves surrounding the blood vessels leading to the kidneys are overactive, which may cause blood pressure to increase. Renal denervation is a procedure where a catheter is placed inside these blood vessels and heat is used to ablate and disable the nerve activity and lower blood pressure.

Hypertension patients that meet the study eligibility criteria will undergo the ultrasound renal denervation procedure using the Paradise System and will be asked to measure their blood pressure throughout the study, including measuring BP out of the clinic setting using a home BP monitoring device provided by the study. Participants will also be asked to answer some questions about their quality of life, health, sleep and emotions. Additional demographic data, medical history and socio-economic data may also be collected. As part of study participation, everyone who receives ultrasound renal denervation will be seen by the study doctor and designated study team members for 60 months (5 years) following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated study informed consent
* Documented history of hypertension
* Documented history of prior or current antihypertensive medication(s)
* Mean seated office systolic BP at screening ≥ 140 mmHg
* Mean pre-procedure home systolic BP of ≥ 135 mmHg
* Estimated glomerular filtration rate (eGFR) of ≥30 mL/min/m2

RADIANCE CAP patients must provide signed and dated informed consent for inclusion in long-term follow-up. No other criteria are required for inclusion.

Exclusion Criteria:

Patients who meet the following will be excluded from participation:

* Patient lacks appropriate renal anatomy for any treatment with the Paradise Catheter
* Patient under the age of 18 years old at the time of consent
* Patient is pregnant
* Patients with transplanted kidney
* Presence of abnormal kidney (or secreting adrenal) tumors

To confirm eligibility for treatment with the Paradise System, the following contraindications listed in the IFU may be determined at the time of procedure prior to treatment:

* Renal arteries with diameter < 3mm and > 8mm
* Renal artery with fibromuscular dysplasia (FMD)
* Stented renal artery
* Renal artery aneurysm
* Renal artery diameter stenosis >30%
* Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension patients in whom lifestyle modifications and antihypertensive medications do not adequately control BP will be identified from the general population by the enrolling center.
  Subjects enrolled in the RADIANCE CAP study will be transferred to the US GPS study after completion of their 12-month follow-up visit in the RADIANCE CAP study, to complete the remainder of the long-term annual follow-up visits under the post approval study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Co-Primary Endpoint #1: Group Mean BP reduction | Baseline to 3-months post-procedure
  * Ho: Reduction in mean home systolic BP from baseline to 3 months < 5 mmHg
  * Ha: Reduction in mean home systolic BP from baseline to 3 months ≥ 5 mmHg
Co-Primary Endpoint #2: Subject Responder | Baseline to 3-months post-procedure
  A subject will be defined as a responder if they achieve any of the following:
  * Control in home BP (defined as systolic BP <130 mmHg) at 3 months and/or
  * Absolute reduction in home systolic BP fall ≥ 5 mmHg at 3 months and/or
  * Reduction in medication burden measured using defined daily dose (DDD)

SECONDARY OUTCOMES:
Change in mean home systolic/diastolic BP in mmHg | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Change in mean office systolic/diastolic BP in mmHg | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Change in home and office pulse pressure | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Change in the number and/or dosage and/or type of antihypertensive medications taken | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Change in patient reported outcomes | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Percentage of patients who are controlled as measured by various cut points of home BP (control to be assessed as both < 130 mmHg systolic and <135 mmHg systolic) office BP (control to also be assessed as <130 mmHg and <140 mmHg systolic) | [baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months]
Percentage of patients who demonstrate a reduction in home systolic BP of ≥ 5mmHg, ≥ 10 mmHg and ≥ 15 mmHg | [at 3, 6, 12, 24, 36, 48 and 60 months compared to baseline]
Percentage of patients who demonstrate a reduction in office systolic BP of ≥ 5mmHg, ≥ 10 mmHg and ≥ 15 mmHg | [at 3, 6, 12, 24, 36, 48 and 60 months compared to baseline]
Change in home and office heart rate | [at 3, 6, 12, 24, 36, 48 and 60 months compared to baseline]

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Sutter Institute for Medical Research, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Rocky Mountain Regional VAMC, Aurora, Colorado
  - Bridgeport Hosptial, Bridgeport, Connecticut
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - University of Miami Health System, Miami, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Southern Illinois University, Memorial Medical Center, Springfield, Illinois
  - Ascension via Christi St. Francis, Wichita, Kansas
  - Touro Infirmary, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Virtua Health, Marlton, New Jersey
  - Albany Medical Center, Albany, New York
  - University at Buffalo, Buffalo, New York
  - NYU Langone Health - Bellevue Hosptial, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Durham VA Health System, Durham, North Carolina
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Ascension Saint Thomas, Nashville, Tennessee
  - Ascension Seton, Austin, Texas
  - Dallas VAMC, Dallas, Texas
  - TCR Institute, Kingwood, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington